CLINICAL TRIAL: NCT04414150
Title: Tolerability, Safety and Pharmacokinetic Characteristics of SHR-1802 in Patients With Advanced Malignancy: a Phase I Clinical Study
Brief Title: A Trial of SHR-1802 in Patients With Failure of Standard Treatment for Advanced Malignant Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1802-I-101
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-06

CONDITIONS: Malignant Tumours
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1802 (Experimental)
  Interventions: Drug: SHR-1802

INTERVENTIONS:
Drug: SHR-1802 — This study will evaluate the preliminary safety, tolerability, pharmacokinetic characteristics and initial efficacy of SHR-1802 The goal is to establish the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of sequential escalating doses of SHR-1802 when administered to patients with locally advanced/ unresectable or metastatic malignant tumours that are refractory to available therapy or for which no standard therapy is available.

SUMMARY:
This is the first study to test SHR-1802 in humans. The primary purpose of this study is to see if SHR-1802 is safe and tolerable for patients with locally advanced/unresectable or metastatic malignancies that are refractory to available therapy or for which no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. Aged 18-75 years (inclusive), males and females;
3. Patient must have histologically or clinically confirmed advanced and/or metastatic malignancies for which failure of standard treatment or lack of effective standard treatment;
4. At least one measurable lesion according to RECIST v1.1;
5. ECOG score of 0-1;
6. Expected survival ≥ 12 weeks;
7. Adequate bone marrow reserve and organ function were confirmed by baseline examination
8. For female patients of childbearing potential or male patients with partners of childbearing potential who are not sterilized by surgical operations, they are required to use a medically approved contraceptive measure during the study treatment period and within 3 months after the end of the study treatment; For female patients of childbearing potential who are not sterilized by surgical operations, they must have a negative serum HCG test result within 72 h prior to study enrollment; and they must not be in the lactation period;

Exclusion Criteria:

1. The presence of any active, known, or suspected autoimmune disease. Type 1 diabetes, which was admitted to receive stable dose of insulin, hypothyroidism, which required only hormone replacement therapy, skin disease with no need to systemic treatment and no acute exacerbation within 1 year before the screening period;
2. Subjects who had received systemic treatment with corticosteroids or other immunosuppressive agents within 28 days prior to initial administration.
3. Known and untreated central nervous system (CNS) or leptomeningeal metastases;
4. Uncontrolled pleural effusion,or ascites requiring recurrent drainage procedures;
5. Uncontrolled cardiac diseases or symptoms;
6. Known hereditary or acquired bleeding and thrombotic tendencies;
7. Patients who have previously received chemotherapy, radiotherapy or surgery which ended within 4 weeks prior to the start of this study; oral molecular targeted therapy with < 5 drug half-lives from the first study dose; or patients with AEs caused by previous treatment (except for alopecia) that have not returned to CTCAE Grade ≤ 1;
8. Known active infection,;
9. Congenital and acquired immune deficiency;
10. HBsAg-positive and HBV DNA > 2000 IU/mL(or 104 copies/mL); HCV RNA copies > ULN;
11. Patients with other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, or family or social factors that could affect the safety of the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Days 1-21

SECONDARY OUTCOMES:
Percentage of patients with adverse events | from the first drug administration to within 90 days for the last SHR-1802 dose
Rates of dose suspension, dose reduction and dose discontinuation caused by investigational drug related adverse events | At pre-defined intervals from initial dose up to 24 months
ORR | At pre-defined intervals from initial dose up to 24 months
DOR | At pre-defined intervals from initial dose up to 24 months
DCR | At pre-defined intervals from initial dose up to 24 months
PFS | At pre-defined intervals from initial dose up to 24 months
Maximum Concentration (Cmax) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Time of Maximum Concentration (Tmax) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Area Under the Curve (AUC) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Terminal Half-Life (T1/2) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Clearance (CL) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Volume of Distribution at Steady State (Vss) of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Evaluation of the immunogenicity of SHR-1802 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
  Serum sampling to assess the potential for anti-drug antibody (ADA) formation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Deng T, Liu Z, Han Z, Zhou H, Liu R, Li Y, Li S, Xiu P, Wang S, Zhang Y, Ba Y. Safety, tolerability, and pharmacokinetics of an anti-LAG-3 antibody SHR-1802 in patients with advanced solid tumors: a phase I dose-escalation and dose-expansion study. Ther Adv Med Oncol. 2023 Jul 29;15:17588359231186025. doi: 10.1177/17588359231186025. eCollection 2023. PMID 37529157